CLINICAL TRIAL: NCT02995811
Title: Characterising Changes in Muscle Quantity and Quality in Patients Requiring Extracorporeal Membrane Oxygen During Critical Illness: 'ECMO-Ultrasound', An Observational Cohort Study
Brief Title: Characterising Changes in Muscle Quantity and Quality in Patients Requiring ECMO Oxygen During Critical Illness
Acronym: ECMO USS
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Euro-ELSO (Unknown)
Responsible Party: Sponsor
Other Study IDs: 208134
Record Dates: First submitted 2016-11-24; First posted 2016-12-16 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Intensive Care Units; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational Cohort: * On Days 1, 3, 7 and 10 of ICU admission, patients will undergo ultrasound assessment of the diaphragm, transverse and rectus abdominis, quadriceps rectus femoris, and tibialis anterior muscles. Imaging all four muscles together requires approximately 1 hour.
  * Physical activity monitoring: On Days 1-10 of ICU admission patients will wear an activity monitor. These devices use several inertial motion sensors to track the movement and acceleration of the limbs in horizontal and vertical directions.
  * Patients will also undergo daily assessment of global peripheral skeletal muscle strength assessed by the Medical Research Council Sum-score and global function measured by the Chelsea Critical Care Physical Assessment Scale
  Interventions: Other: Observational Cohort

INTERVENTIONS:
Other: Observational Cohort — Ultrasound assessment of 4 muscles, activity monitoring, daily global peripheral skeletal muscle strength

SUMMARY:
This study will identify the changes in different muscles of patients receiving Extracorporeal Membrane Oxygenation (ECMO) during critical illness and admission to Intensive Care Unit (ICU). The information will help guide development of treatments such as exercise that may help to reduce the amount of muscle wasting that can occur during critical illness.

DETAILED DESCRIPTION:
Admission to the intensive care unit (ICU) with critical illness is typically associated with profound physical impairments including peripheral skeletal muscle wasting and dysfunction. These effects demonstrate a rapid onset from the point of ICU admission, affect those with higher illness acuity to greater levels, and contribute to the development of intensive care unit-acquired weakness (ICU-AW) defined as severe upper and lower limb muscle weakness.

Muscle structure has traditionally been evaluated using complex scanning approaches such as computed tomography or dual energy x-ray absorptiometry, however there are a number of caveats to their use in the clinical environment of critical care. Ionising radiation involved precludes their use in large populations, and especially for performance of sequential measurements. Whilst magnetic resonance imaging avoids this concern, practical limitations exist around scanning time and accessibility. In addition, all these imaging modalities require transfer out of the ICU environment, further restricting their application to acutely unwell, unstable patients. Finally, in addition to their expense, the nature of imaging using these approaches means that only a limited number of muscles may be assessed at any one time.

Ultrasound has emerged in recent years as a technique with significant clinical utility for assessing and monitoring the trajectory of change in muscle during acute critical illness. A range of parameters of muscle architecture and quality can be measured and data from the critical illness population is growing. Advantages of ultrasound include feasibility of bedside assessment, and that is it non-ionising, non-invasive and effort-independent with equipment is readily available in the critical care environment. Ultrasound imaging has robust clinimetric properties and predictive utility for morbidity and other clinical endpoints including mortality and hospital readmission.

A number of observational cohort studies have conducted sequential measurements of a range of respiratory and peripheral skeletal muscle groups during critical illness, characterising the decline in both muscle quantity and quality as a result of the acute insult. However no studies to date have included assessment of the abdominal muscles in critically ill patients necessary for core stability, trunk control and postural maintenance and therefore of significant clinical importance during the rehabilitation process.

In addition, whilst hypoxia has been found to be associated with greater muscle attenuation, no study has examined the relative changes in muscle in patients receiving extracorporeal membrane oxygenation (ECMO). ECMO is a ventilator support therapy primarily delivered to critically ill patients with severe respiratory failure where the hypoxic state is corrected.

The aim of this study is therefore to characterise sequential changes across respiratory, trunk and peripheral skeletal muscles in critically ill patients requiring ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Adult, ≥18years
* Requiring ECMO for management of severe respiratory failure
* Likely to remain in the ICU for 10days

Exclusion Criteria:

* Pregnancy
* Neurological injury e.g. stroke, acquired brain injury
* Trauma injury e.g. amputation, multiple fractures
* Clinical presentation precluding ultrasound imaging of muscle at the time of assessment
* Not expected to survive more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted to the ICU with critical illness requiring ECMO
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Sequential changes in parameters of muscle architecture of the muscles in critically ill patients requiring ECMO by Ultrasound | 10 days
Sequential changes in quality of the muscles in critically ill patients requiring ECMO by Ultrasound | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Barrett, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data